CLINICAL TRIAL: NCT06038448
Title: Efficacy of Reduction of the Balloon Volume for Prevention of Postoperative Catheter-related Bladder Discomfort in Patients Undergoing Non-lower Urinary Tract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TCRD112-017
Record Dates: First submitted 2023-09-08; First posted 2023-09-14 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-05

CONDITIONS: Catheter-Related Bladder Discomfort; Urinary Catheter
Keywords: urinary catheter; Catheter-Related Bladder Discomfort; balloon; nursing

STUDY DESIGN:
Intervention Model Description: parallel into two groups, each urinary catheter balloon size 10mL and 5mL
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effect of normal 10ml balloon volume on postoperative CRBD in non-LUTS patients (Active Comparator): Efficacy of normal 10ml balloon volume for prevention of postoperative catheter-related bladder discomfort in patients undergoing non-lower urinary tract surgery
  Interventions: Procedure: Urinary catheter balloon size
- Effect of reduction of 5ml balloon volume for postoperative CRBD in patients undergoing non-LUTS (Active Comparator): Efficacy of reduction of 5ml the balloon volume for prevention of postoperative catheter-related bladder discomfort in patients undergoing non-lower urinary tract surgery
  Interventions: Procedure: Urinary catheter balloon size

INTERVENTIONS:
Procedure: Urinary catheter balloon size — The investigators will collect 120 participants divided into two groups ,in different procedure(stone procedure, herniarraphy, nephrectomy), and the investigators used different urinary catheter balloon size(10ml and 5ml), tp investigate the patient with the severity of catheter-related bladder discomfort.

SUMMARY:
CRBD is related to different degrees of irritation caused by the volume of the balloon in the urinary catheter, and when CRBD occurs, it may cause severe postoperative pain and trauma by self-removal of the catheter, further leading complications. Although many drugs can improve CRBD, measures that can be immediately intervened by non-nursing staff at any time and even have different side effects on patients due to drug use.Therefore, the author wants to use this study to explore the reduction of catheter balloon volume can effectively reduce the degree of CRBD, is a non-invasive and immediately executable nursing treatment.the quality of clinical care and hospitalization of the patient can be further improved, reducing the patient's inappropriate, thereby improving the quality of medical care.

DETAILED DESCRIPTION:
Catheter-Related Bladder Discomfort (CRBD) has been attached importance in recent years. Reducing the discomfort of patients with effective treatment is a part of our medical and nursing care that needs to be paid more attention to. The literature has pointed out that CRBD is related to different degrees of irritation caused by the volume of the balloon in the urinary catheter, and when CRBD occurs, it may cause severe postoperative pain and trauma by self-removal of the catheter, further leading to urethral injury and subsequent urethral stricture, and complications such as bleeding, surgical wound dehiscence, and arrhythmia. Although many drugs can improve CRBD, measures that can be immediately intervened by non-nursing staff at any time and even have different side effects on patients due to drug use.

In the past 20 years, only one piece of literature has discussed the effect of catheter balloon volume on CRBD, and the sample size is relatively small and even not related to the Asian region. Therefore, the author wants to use this study to explore the reduction of catheter balloon volume can effectively reduce the degree of CRBD, the investigators will collect in different procedure(stone procedure, herniarraphy, nephrectomy), and the investigators used different urinary catheter balloon size(10ml and 5ml), tp investigate the patient with the severity of catheter-related bladder discomfort.In addition to reducing the side effects of patients due to drug use, is a non-invasive and immediately executable nursing treatment.

Further, if post-evidence nursing intervention can effectively reduce the CRBD generated, thereby increasing the patient's comfort, and allowing the patient to cooperate more with the treatment to achieve an effective therapeutic effect, thereby improving the quality of care and the enlargement of recovery.

Eventually, the quality of clinical care and hospitalization of the patient can be further improved, reducing the patient's inappropriate, thereby improving the quality of medical care.

Key words: Catheter-Related Bladder Discomfort, urinary catheter, balloon, nursing

ELIGIBILITY:
Inclusion Criteria:

* age from 20-80 year-old
* in urological surgery under the general anesthesia
* 2 arms: (1)non-lower urinary tract surgery: hernia, and nephrectomy surgery , (2) lower urinary tract surgery: stone surgery after ureter catheter insertion.

Exclusion Criteria:

* Patients not undergoing hernia repair or nephrectomy.
* Patients who are not undergoing ureteral lithotripsy and renal stone extraction.
* Those who are already using drugs for overactive bladder or prostatic hypertrophy.
* Retrograde intrarenal surgery (RIRS) for stone extraction.
* People with dementia.
* Patients with cognitive impairment.
* Patients with impaired consciousness.
* Patients who are unable to communicate verbally.
* The subject had participated in other experimental drug trials one month before the study entered.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-18 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Degree of Catheter-related Bladder Discomfort | Return to the ward after surgery 0 hours.3 hours.12 hours
  Likert scale 0.1.2.3,the minimum value is 0 and the maximum value is 3. The larger the number, the more serious the discomfort is.

SECONDARY OUTCOMES:
Visual analog scale for pain severity | Return to the ward after surgery 0 hours.3 hours.12 hours
  0 to 10,the minimum value is 0 and the maximum value is 10. The larger the number, the more serious the discomfort is.

IPD SHARING:
Plan to Share IPD: No